CLINICAL TRIAL: NCT05248321
Title: Precise Application of Topical Tranexamic Acid to Enhance Endoscopic Hemostasis for Peptic Ulcer Bleeding: A Randomized Controlled Study
Brief Title: Precise Delivery of Tranexamic Acid to Enhance Endoscopic Hemostasis for Peptic Ulcer Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-BR-110-085
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Peptic Ulcer Hemorrhage
Keywords: Peptic ulcer; Tranexamic acid powder spray; Recurrent ulcer bleeding
MeSH Terms: conditions — Peptic Ulcer Hemorrhage; Peptic Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extra treatment (ET) group (Experimental): In the extra treatment (ET) group, standard endoscopic therapy will be performed to the bleeding peptic ulcer by local injection of diluted epinephrine 1:10 000 in combination with either heater probe coagulation, hemoclipping and/or rubber band ligation. Afterwards, we will apply 1.25g tranexamic acid powder via the endoscopy to the peptic ulcer before the end of endoscopic exam. After the first endoscopy, the patient will receive a 3-day continuous high-dose (8 mg/h) PPI infusion and Rockall score assessment as current guideline's recommendation. In patients with Rockall scores ≥6, after 3-day intravenous PPI infusion, we will apply oral twice-daily PPI for 11 days followed by once-daily PPI after then. In patients with Rockall scores <6, we will apply once-daily PPI after 3-day intravenous PPI infusion. A second-look esophagogastroduodenoscopy (EGD) will be performed 2-3 days after the initial endoscopy, aiming to survey if major SRH of peptic ulcer persists.
  Interventions: Drug: Tranexamic Acid Powder
- standard treatment (ST) group (No Intervention): In the standard treatment (ST) group, the endoscopic exam ends after standard endoscopic therapy. After the first endoscopy, the patient will receive a 3-day continuous high-dose (8 mg/h) PPI infusion and Rockall score assessment as current guideline's recommendation. In patients with Rockall scores ≥6, after 3-day intravenous PPI infusion, we will apply oral twice-daily PPI for 11 days followed by once-daily PPI after then. In patients with Rockall scores <6, we will apply once-daily PPI after 3-day intravenous PPI infusion. A second-look esophagogastroduodenoscopy (EGD) will be performed 2-3 days after the initial endoscopy, aiming to survey if major SRH of peptic ulcer persists.

INTERVENTIONS:
Drug: Tranexamic Acid Powder — 2g tranexamic acid powder will be given via the endoscopy directly to the peptic ulcer
  Other Names: Tranexamic acid powder spray from endoscopy
  Arms: Extra treatment (ET) group

SUMMARY:
Peptic ulcer bleeding is a common emergency for patients who need therapeutic endoscopy. According to international guidelines and Taiwan consensus, the standard therapy included proton pump inhibitor (PPI) and endoscopic therapy. For high-risk peptic ulcers, such as active spurting, oozing bleeding, a nonbleeding visible vessel or ulcers with adherent clots, we apply endoscopic hemostasis with epinephrine injection in combination with either heater probe coagulation, hemoclipping and/or rubber band ligation. Parenteral high-dose PPI is administered after endoscopic hemostasis. Though current standard endoscopic therapy plus PPI infusion are highly effective, 5%-10% of the patients still experience recurrence of bleeding after the initial treatment. It is still an important issue to reduce recurrent peptic ulcer bleeding after standard endoscopic therapy.

Tranexamic acid reduces bleeding by inhibiting clot breakdown by inhibiting the degradation of fibrin by plasmin. It is effective to be used topically to reduce bleeding during surgery. However, the effect of application of tranexamic acid orally or intravenously for gastrointestinal bleeding was still controversial, probably because that the route of tranexamic acid use is not precise at the bleeding site. Tranexamic acid has anti-fibrinolytic effects at the bleeding site, so it is possible that use of tranexamic acid locally may have better efficacy than via intravenous or oral route. We propose to investigate the effectiveness and safety when using tranexamic acid locally under endoscopic guidance in patients with peptic ulcer bleeding after standard endoscopic therapy.

DETAILED DESCRIPTION:
Upper gastrointestinal (UGI) hemorrhage is a common emergency for patients who need therapeutic endoscopy. Among these patients, peptic ulcer bleeding is the most common causes in UGI bleeding with risk for mortality. According to Taiwan consensus, standard therapy included proton pump inhibitor (PPI) and endoscopic therapy. We use Rockall score and Forrest classification to decide the use of endoscopic therapy and predict recurrent bleeding rate of the peptic ulcer. For high-risk peptic ulcer, such as active spurting (Forrest classification Ia), oozing bleeding (Forrest classification Ib), a nonbleeding visible vessel (Forrest classification IIa) or ulcers with adherent clots (Forrest classification IIb), we apply endoscopic hemostasis with epinephrine injection in combination with either heater probe coagulation, hemoclipping and/or rubber band ligation. Standard endoscopic hemostasis is highly effective, with overall success rates of 85%-95% in stopping hemorrhage. However, 5%-10% of the patients still experience recurrence of bleeding after the initial endoscopic hemostasis, especially in those with Rockall scores≥6. Although most patients with peptic ulcer bleeding can be treated successfully via standard endoscopic therapy and PPI use, some patients suffered from continuous bleeding or recurrent bleeding later after therapeutic endoscopy according to our previous studies. It is still an important issue to reduce recurrent peptic ulcer bleeding after standard endoscopic therapy.

Previous studies have shown tranexamic acid as a well-known antifibrinolytic agents. Tranexamic acid reduces bleeding by inhibiting clot breakdown by inhibiting the degradation of fibrin by plasmin. Tranexamic acid has been proved to reduces blood loss in patients with surgical bleeding, the need for transfusion, and reduce mortality due to traumatic bleeding. It can also be used topically to reduce bleeding. Application of tranexamic acid for gastrointestinal bleeding was still controversial. HALT-IT trial showed that intravenous tranexamic acid did not reduce death from gastrointestinal bleeding. We assume the ineffectiveness of tranexamic acid may due to intravenous use rather than local use precisely at the bleeding site. The role of endoscopic local administration of antifibrinolytic agents remains unclear. Tranexamic acid has anti-fibrinolytic effects in bleeding site, so it is reasonable that local use of tranexamic acid may have stronger efficacy than intravenous use.

We propose to investigate the effectiveness and safety when using tranexamic acid locally under endoscopic guidance in patients with peptic ulcer bleeding after standard endoscopic therapy. This is an important issue because there are many patients with recurrent GI bleeding who suffered from potential risk of death. We apply tranexamic acid to the precise bleeding site, and anticipate that we can have better outcome for those patients.

Subjects and protocols Participants will be recruited from the volunteers with peptic bleeding in National Cheng Kung University Hospital. Eligible participants included patients aged ≥20 years who will accept esophagogastroduodenoscopy (EGD) for melena, hematochezia, hematemesis or coffee-ground fluid or bloody fluid drained from nasogastric tube. Patient consent form will be given to all patients before EGD. The participants will receive endoscopic survey, and we will enroll patients with peptic ulcer with major stigmata of recent hemorrhage. Major stigmata of recent hemorrhage (SRH) include active spurting (Forrest classification Ia), oozing bleeding (Forrest classification Ib), a nonbleeding visible vessel (Forrest classification IIa) or ulcers with adherent clots (Forrest classification IIb). Exclusion criteria includes poor renal function (serum creatinine > 2.9mg/dL), tumor ulcer bleeding, allergy to tranexamic acid, whose antiplatelet agent/anticoagulation agent could not be transiently withdrawn. We will apply standard endoscopic therapy to the bleeding peptic ulcer by local injection of diluted epinephrine 1:10 000 in combination with either heater probe coagulation, hemoclipping and/or rubber band ligation. After then, we will assign the patient to either standard therapy (ST) group or extra therapy (ET) group following block randomization procedures with a 1:1 allocation ratio. Balanced combinations of equal number for the two groups were within the blocks. Blocks are then randomly chosen to determine the patients' assignment into the two groups. The allocation sequence was concealed until the researchers had randomized the patients. In the standard treatment (ST) group, the endoscopic exam ends after standard endoscopic therapy as mentioned above. In the extra treatment (ET) group, we will apply 1.25g tranexamic acid powder via the endoscopy to the peptic ulcer before the end of endoscopic exam. Both groups then receive a 3-day continuous high-dose (8 mg/h) PPI infusion and Rockall score assessment as current guideline's recommendation. In patients with Rockall scores ≥6, after 3-day intravenous PPI infusion, we will apply oral twice-daily PPI for 11 days followed by once-daily PPI after then. In patients with Rockall scores <6, we will apply once-daily PPI after 3-day intravenous PPI infusion. A second-look esophagogastroduodenoscopy (EGD) will be performed 2-3 days after the initial endoscopy, aiming to survey if major SRH of peptic ulcer persists.

All enrolled patients were included in the final analysis. The patients' underlying medical disease and medication will be reviewed. For patients who received antiplatelet therapy for prophylaxis of established cardiovascular or cerebrovascular diseases, the treatment was discontinued for 3 days after EGD. The antiplatelet therapy was resumed with clopidogrel 75 mg/day or aspirin 100 mg/day on the 4th day.

Blood tests Blood sample is obtained to measure blood urine nitrogen, creatinine, albumin, total bilirubin, hemoglobin, platelet, prothrombin time (PT) and activated partial thromboplastin time (APTT). All lab data are checked by central laboratory of National Cheng Kung University Hospital.

Outcome measures All patients will be monitored for 28 days after the first EGD. The primary end point is the early treatment failure within 4 days. Early treatment failure was defined as (1) continuous melena, hematochezia, bloody drainage from a nasogastric tube, hemodynamic instability (systolic blood pressure <90 mm Hg, heart rate >120 bpm), or a drop in serum hemoglobin >2 g/dL with the subsequent EGD confirmation of index ulcer with major SRH, or (2) index ulcer with major SRH in need of repeated endoscopic hemostasis during the second-look EGD. For each patient with suspected rebleeding, we will perform an EGD to confirm any blood or coffee-ground materials in the stomach, or the persistence of stigmata indicating recent hemorrhage. The EGD also determines whether the source of rebleeding is the peptic ulcer or other non-ulcer bleeding source. The secondary outcomes included (1) rebleeding from the index ulcer within 28 days, (2) index ulcer rebleeding requiring transarterial embolization (TAE) or emergent surgery; (3) length of hospitalization; (4) PRBC transfusion units, (5) mortality; (6) severe adverse events from tranexamic acid, e.g., seizures and thromboembolic events.

Statistical analysis The pilot study will enroll total sixty cases, including 30 cases in the ST group and 30 cases in the ET group, respectively. Data related to baseline characteristics and end points were evaluated using the Student t test, Pearson's χ2 test or Fisher's exact test and the Mann-Whitney U test. In the survival analysis, the log-rank test was used to compare the Kaplan-Meier curves among the two study groups. All tests were two-tailed and p values <0.05 indicated significant differences.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peptic ulcer with major stigmata of recent hemorrhage receiving EGD therapy

Exclusion Criteria:

* Poor renal function (serum creatinine > 2.9mg/dL)
* Tumor ulcer bleeding
* Patients allergy to tranexamic acid
* Whose antiplatelet agent/anticoagulation agent could not be transiently withdrawn

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Rate of the early treatment failure of the index ulcer | 4 days
  We monitor if early treatment failure of the peptic ulcer occurs after the first endoscopic therapy within 4 days. Early treatment failure was defined as (1) continuous melena, hematochezia, bloody drainage from a nasogastric tube, hemodynamic instability (systolic blood pressure <90 mm Hg, heart rate >120 bpm), or a drop in serum hemoglobin >2 g/dL with the subsequent EGD confirmation of index ulcer with major SRH, or (2) index ulcer with major SRH in need of repeated endoscopic hemostasis during the second-look EGD.

SECONDARY OUTCOMES:
Rate of the recurrent bleeding from the index ulcer | 28 days
  We monitor if rebleeding of the peptic ulcer occurs.
PRBC transfusion units | 28 days
  The total units of PRBC transfusion during the hostpital stays
The length of hospitalization | 28 days
  We record the total days of hospitalization.
Recurrent ulcer bleeding requiring transarterial embolization or emergent surgery | 28 days
  We record if recurrent ulcer bleeding occurs and require hemostasis by emergent transarterial embolization or emergent surgery.
The mortality | 28 days
  We record all-cause mortality after the first EGD within 28 days.
The severe adverse events from tranexamic acid powder | 28 days
  The severe adverse effects includes seizures and thromboembolic events.

CONTACTS AND LOCATIONS:
Overall Officials: Xi-Zhang Lin, M.D., Study Chair — National Cheng-Kung University Hospital
Locations (1):
- National Cheng-Kung University Hospital, Tainan, NONE Selected, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Result] Yavorski RT, Wong RK, Maydonovitch C, Battin LS, Furnia A, Amundson DE. Analysis of 3,294 cases of upper gastrointestinal bleeding in military medical facilities. Am J Gastroenterol. 1995 Apr;90(4):568-73. PMID 7717312
- [Result] Sheu BS, Wu CY, Wu MS, Chiu CT, Lin CC, Hsu PI, Cheng HC, Lee TY, Wang HP, Lin JT. Consensus on control of risky nonvariceal upper gastrointestinal bleeding in Taiwan with National Health Insurance. Biomed Res Int. 2014;2014:563707. doi: 10.1155/2014/563707. Epub 2014 Aug 14. PMID 25197649
- [Result] Yang EH, Wu CT, Kuo HY, Chen WY, Sheu BS, Cheng HC. The recurrent bleeding risk of a Forrest IIc lesion at the second-look endoscopy can be indicated by high Rockall scores >/= 6. Surg Endosc. 2020 Apr;34(4):1592-1601. doi: 10.1007/s00464-019-06919-3. Epub 2019 Jun 20. PMID 31222633
- [Result] Gralnek IM, Dumonceau JM, Kuipers EJ, Lanas A, Sanders DS, Kurien M, Rotondano G, Hucl T, Dinis-Ribeiro M, Marmo R, Racz I, Arezzo A, Hoffmann RT, Lesur G, de Franchis R, Aabakken L, Veitch A, Radaelli F, Salgueiro P, Cardoso R, Maia L, Zullo A, Cipolletta L, Hassan C. Diagnosis and management of nonvariceal upper gastrointestinal hemorrhage: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2015 Oct;47(10):a1-46. doi: 10.1055/s-0034-1393172. Epub 2015 Sep 29. PMID 26417980
- [Result] Lee JH, Kim BK, Seol DC, Byun SJ, Park KH, Sung IK, Park HS, Shim CS. Rescue endoscopic bleeding control for nonvariceal upper gastrointestinal hemorrhage using clipping and detachable snaring. Endoscopy. 2013 Jun;45(6):489-92. doi: 10.1055/s-0032-1326375. Epub 2013 Apr 11. PMID 23580408
- [Result] Yang EH, Cheng HC, Wu CT, Chen WY, Lin MY, Sheu BS. Peptic ulcer bleeding patients with Rockall scores >/=6 are at risk of long-term ulcer rebleeding: A 3.5-year prospective longitudinal study. J Gastroenterol Hepatol. 2018 Jan;33(1):156-163. doi: 10.1111/jgh.13822. PMID 28497645
- [Result] Picetti R, Shakur-Still H, Medcalf RL, Standing JF, Roberts I. What concentration of tranexamic acid is needed to inhibit fibrinolysis? A systematic review of pharmacodynamics studies. Blood Coagul Fibrinolysis. 2019 Jan;30(1):1-10. doi: 10.1097/MBC.0000000000000789. PMID 30585835
- [Result] Hunt BJ. The current place of tranexamic acid in the management of bleeding. Anaesthesia. 2015 Jan;70 Suppl 1:50-3, e18. doi: 10.1111/anae.12910. PMID 25440395
- [Result] Ker K, Beecher D, Roberts I. Topical application of tranexamic acid for the reduction of bleeding. Cochrane Database Syst Rev. 2013 Jul 23;2013(7):CD010562. doi: 10.1002/14651858.CD010562.pub2. PMID 23881695
- [Result] HALT-IT Trial Collaborators. Effects of a high-dose 24-h infusion of tranexamic acid on death and thromboembolic events in patients with acute gastrointestinal bleeding (HALT-IT): an international randomised, double-blind, placebo-controlled trial. Lancet. 2020 Jun 20;395(10241):1927-1936. doi: 10.1016/S0140-6736(20)30848-5. PMID 32563378
- [Result] Cheng HC, Wu CT, Chang WL, Cheng WC, Chen WY, Sheu BS. Double oral esomeprazole after a 3-day intravenous esomeprazole infusion reduces recurrent peptic ulcer bleeding in high-risk patients: a randomised controlled study. Gut. 2014 Dec;63(12):1864-72. doi: 10.1136/gutjnl-2013-306531. Epub 2014 Mar 21. PMID 24658598
- [Derived] Chiang HC, Chen PJ, Yang EH, Hsieh MT, Shih IC, Cheng HC, Chang WL, Chen WY, Chiu HC, Kuo HY, Tsai WC, Lo YN, Yang KC, Chiang CM, Chen WC, Huang KK, Tseng HH, Chen CY, Lin XZ, Chuang CH. Precise application of topical tranexamic acid to enhance endoscopic hemostasis for peptic ulcer bleeding: a randomized controlled study (with video). Gastrointest Endosc. 2023 Nov;98(5):755-764. doi: 10.1016/j.gie.2023.06.013. Epub 2023 Jun 24. PMID 37356632